CLINICAL TRIAL: NCT05287035
Title: Perioperative IV Steroid Administration Lowers Post-operative Pain Levels and Opioid Use in Pediatric Patients After Posterior Spinal Fusion and Instrumentation for Spine Deformity.
Brief Title: Spinal Fusions Steroid Study
Acronym: SFSS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Brian Kaufman, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00002340
Record Dates: First submitted 2022-02-24; First posted 2022-03-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Spinal Fusion
MeSH Terms: interventions — Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: The study will be a double blinded (patient, surgeon) prospective randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patient and surgeon will be masked. Anesthesiologist will not be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Steroid injection (Active Comparator): Dexamethasone will be injected 1 dose intraoperatively, 3 doses post-operatively every 8hrs
  Interventions: Drug: Dexamethasone injection
- Saline solution (Placebo Comparator): Saline will be injected 1 dose intraoperatively, 3 doses post-operatively every 8hrs
  Interventions: Other: Saline injection

INTERVENTIONS:
Drug: Dexamethasone injection — Dexamethasone will be injected at the dosage recommended by the FDA.
  Arms: Steroid injection
Other: Saline injection — Saline will be injected for the placebo arm of the study.
  Arms: Saline solution

SUMMARY:
Current efforts to improve pain alleviation focus on non-opioid pharmaceuticals. Intravenous perioperative corticosteroid administration has been suggested as an alternative method for post-operative pain control. The evidence regarding perioperative intravenous corticosteroids to help alleviate post-operative pain is mixed. Some meta-analyses report decreased opioid consumption and decreased pain intensity after a variety of surgical procedures. However, a study of larger orthopedic procedures found no benefit. The catabolic and immunosuppressant effects of corticosteroids also pose issues with wound healing and infection, which can have severe consequences after spine surgery. There is limited data on the effect of perioperative intravenous steroid administration on pain alleviation in children having surgery to address spine deformity. A recent retrospective review demonstrated that perioperative corticosteroid administration was associated with a statistically significant decrease in opioid medication utilization among children and adolescents after spinal deformity surgery. While not increasing the risk of postoperative complications. The investigators hypothesize that the administration of perioperative intravenous dexamethasone will demonstrate a clinically meaningful and statistically significant decrease in postoperative pain intensity, need for opioid medications, time to ambulation, and length of stay in children recovering from surgery for spine deformity.

ELIGIBILITY:
Inclusion Criteria:

* Meets operative criteria for posterior spinal instrumented fusion for AIS
* Parental consent

Exclusion Criteria:

* Revision procedure
* Other associated conditions which may alter the postoperative course

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Time to initial ambulation post-operatively and distance ambulated in first physical therapy session. | 1 week
  The investigators will assess the time to initial ambulation in reference to the surgical stop time recorded in the chart. This time will be calculated in minutes. The total minutes until first ambulation for both arms of the study will be compared. The investigators will assess measure, in feet, the distance patients ambulate during the initial session with physical therapy postoperatively. The distance, in feet, ambulated by patient in each arm of the study will be directly compared.
Length of stay in hospital | 1 week
  The investigators will measure the number of days in the hospital from the date of surgery
Morphine equivalents use | 1 week
  The investigators will record the amount of morphine equivalents utilized by patients in the post-operative in-hospital period to compare the use of intravenous narcotics in a quantifiable fashion between the two study groups.

SECONDARY OUTCOMES:
Return to emergency department | 12 months
  The investigators will track rates of return to the Emergency Department and/or return for hospital admission after discharge from the hospital. Rates of return to the Emergency Department and/or need for hospital admission will be stratified across 30 day, 90 day, and 365 day intervals after discharge from the hospital. Additionally, data will be collected by the investigators on the cause of return to the Emergency Department and/or return for hospital admission. Examples of cause for return will include: insufficient pain control at home, concerning neurologic findings, inability to tolerate per os nutrition, inability to urinate or defecate, wound dehiscence or drainage, and all other causes.
  We will keep track of patients that need to return to the emergency department for any reason.
Return to school | 3 months
  The investigators will determine the length of time it takes a patient to return to school after surgery.
Pain score at discharge | 1 week
  The investigators will record the patient's pain score at regular intervals during hospital admission (typically assessed every 4 hours by the nursing staff) as well as recording pain score at time of discharge from the hospital. Pain scores will be recorded in two fashions. Primarily, a pain score of 0 to 10 will be recorded whereby a patient-reported score of "0" indicates no perceived pain and a score of "10" would indicate severe and intractable pain. Secondarily, as this study involves pediatric patients, the investigators will record pain using the Wong-Baker FACES Pain Rating Scale that similarly uses a scoring system of 0 to 10, but additionally includes illustrations of faces to guide pediatric patients in relating their pain to a numeric score. The Wong-Baker FACES Pain Rating Scale is a validated tool for recording pain levels in pediatric patients and is widely used within the investigators hospital system.

CONTACTS AND LOCATIONS:
Locations (1):
- Dell Children's Medical Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We plan to publish the results of this study. All protected health information (PHI) will be delinked from the participant and will only be accessed by authorized research personnel. IPD will be destroyed at the end of the study.

REFERENCES:
- [Result] Sinatra RS, Torres J, Bustos AM. Pain management after major orthopaedic surgery: current strategies and new concepts. J Am Acad Orthop Surg. 2002 Mar-Apr;10(2):117-29. doi: 10.5435/00124635-200203000-00007. PMID 11929206
- [Result] Fletcher ND, Ruska T, Austin TM, Guisse NF, Murphy JS, Bruce RW Jr. Postoperative Dexamethasone Following Posterior Spinal Fusion for Adolescent Idiopathic Scoliosis. J Bone Joint Surg Am. 2020 Oct 21;102(20):1807-1813. doi: 10.2106/JBJS.20.00259. PMID 33086348
- [Result] Pobereskin LH, Sneyd JR. Does wound irrigation with triamcinolone reduce pain after surgery to the lumbar spine? Br J Anaesth. 2000 Jun;84(6):731-4. doi: 10.1093/oxfordjournals.bja.a013583. PMID 10895746
- [Result] Jirarattanaphochai K, Jung S, Thienthong S, Krisanaprakornkit W, Sumananont C. Peridural methylprednisolone and wound infiltration with bupivacaine for postoperative pain control after posterior lumbar spine surgery: a randomized double-blinded placebo-controlled trial. Spine (Phila Pa 1976). 2007 Mar 15;32(6):609-16; discussion 617. doi: 10.1097/01.brs.0000257541.91728.a1. PMID 17413463
- [Result] Wittayapairoj A, Wittayapairoj K, Kulawong A, Huntula Y. Effect of intermediate dose dexamethasone on post-operative pain in lumbar spine surgery: A randomized, triple-blind, placebo-controlled trial. Asian J Anesthesiol. 2017 Sep;55(3):73-77. doi: 10.1016/j.aja.2017.08.001. Epub 2017 Sep 18. PMID 28986051
- [Result] Sharma M, Gupta S, Purohit S, Goyal AK. The Effect of Intravenous Dexamethasone on Intraoperative and Early Postoperative Pain in Lumbar Spine Surgery: A Randomized Double-Blind Placebo-Controlled Study. Anesth Essays Res. 2018 Oct-Dec;12(4):803-808. doi: 10.4103/aer.AER_115_18. PMID 30662111
- [Result] Hernandez-Palazon J, Tortosa JA, Martinez-Lage JF, Perez-Flores D. Intravenous administration of propacetamol reduces morphine consumption after spinal fusion surgery. Anesth Analg. 2001 Jun;92(6):1473-6. doi: 10.1097/00000539-200106000-00024. PMID 11375828
- [Result] Fletcher ND, Shourbaji N, Mitchell PM, Oswald TS, Devito DP, Bruce RW. Clinical and economic implications of early discharge following posterior spinal fusion for adolescent idiopathic scoliosis. J Child Orthop. 2014 May;8(3):257-63. doi: 10.1007/s11832-014-0587-y. Epub 2014 Apr 27. PMID 24770995
- [Result] Munro HM, Walton SR, Malviya S, Merkel S, Voepel-Lewis T, Loder RT, Farley FA. Low-dose ketorolac improves analgesia and reduces morphine requirements following posterior spinal fusion in adolescents. Can J Anaesth. 2002 May;49(5):461-6. doi: 10.1007/BF03017921. PMID 11983659
- [Result] Lee CS, Merchant S, Chidambaran V. Postoperative Pain Management in Pediatric Spinal Fusion Surgery for Idiopathic Scoliosis. Paediatr Drugs. 2020 Dec;22(6):575-601. doi: 10.1007/s40272-020-00423-1. Epub 2020 Oct 23. PMID 33094437
- [Result] Liu K, Hsu CC, Chia YY. Effect of dexamethasone on postoperative emesis and pain. Br J Anaesth. 1998 Jan;80(1):85-6. doi: 10.1093/bja/80.1.85. PMID 9505784
- [Result] Romundstad L, Breivik H, Niemi G, Helle A, Stubhaug A. Methylprednisolone intravenously 1 day after surgery has sustained analgesic and opioid-sparing effects. Acta Anaesthesiol Scand. 2004 Nov;48(10):1223-31. doi: 10.1111/j.1399-6576.2004.00480.x. PMID 15504180
- [Result] Aasboe V, Raeder JC, Groegaard B. Betamethasone reduces postoperative pain and nausea after ambulatory surgery. Anesth Analg. 1998 Aug;87(2):319-23. doi: 10.1097/00000539-199808000-00015. PMID 9706923
- [Result] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857